CLINICAL TRIAL: NCT00455130
Title: A Phase 2 Study to Determine the Safety and Efficacy of Inhaled Dry Powder Mannitol in Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Syntara (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DPM-CF-201
Record Dates: First submitted 2007-04-02; First posted 2007-04-03 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Cystic Fibrosis
Keywords: mannitol; cystic fibrosis; mucolytic; mucoactive
MeSH Terms: conditions — Cystic Fibrosis

INTERVENTIONS:
Drug: Inhaled mannitol

SUMMARY:
Cystic fibrosis is the most frequent lethal genetic disease of childhood. Causes disruption of glandular function of the pancreas, intestine, liver, lungs (causing chronic lung infection with emphysema), sweat glands and reproductive organs. We know that many CF patients die of lung failure, brought about in part by repeated lung infections caused by thick, sticky mucus that cannot be readily cleared from the lung.

Inhaled mannitol is an osmotic agent that has been investigated in a number of small studies that have examined mucociliary clearance, quality of life and lung function in CF and bronchiectasis. The promising results of these studies warrant futher investigation. The aim of this study is to assess the safety and efficacy of inhaled mannitol when administered twice a day over two weeks in CF.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of cystic fibrosis (sweat test/genotype)
2. Aged 8 years or older
3. Have FEV1 between 40% and 80% of predicted for height, age and gender OR a decrease in FEV1 of 20% or more than that recorded 6-12 months previously.
4. As determined by the investigator, are capable and willing to

   * Use the study diary as required for this protocol
   * Able to perform all of the techniques necessary to measure lung function
   * Able to administer the dry powder mannitol
5. Are capable of and have given informed consent
6. Clinically stable at study entry

Exclusion Criteria:

1. Investigators, site personnel directly affiliated with this study, and their immediate families.
2. Subjects under the age of 8 years.
3. Subjects with currently active asthma
4. Subjects using hypertonic saline treatment in the last 2 weeks
5. Considered "terminally ill" or listed for transplantation
6. Requiring home oxygen or assisted ventilation
7. Colonisation with Burkholderia cepacia
8. Significant episode of hemoptysis (>60 mls) in the previous 12 months
9. Myocardial Infarction in the six months prior to enrolment.
10. Cerebral Vascular Accident in the six months prior to enrolment.
11. Ocular surgery in the three months prior to enrolment.
12. Abdominal surgery in the three months prior to enrolment.
13. Subjects who are breast feeding or pregnant.
14. Female subjects of reproductive capability, not using a reliable form of contraception
15. Inability to obtain informed consent from the subject or subject's authorised representative.
16. Subjects who have participated in another investigative drug study parallel to, or within 4 weeks of study entry.
17. Known intolerance to mannitol or beta2 agonists.
18. Uncontrolled hypertension - systolic BP > 160 and or diastoli

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-03; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
FEV1

SECONDARY OUTCOMES:
Other measures of lung function
Quality of life
Sputum microbiology
Sputum rheology
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Brett Charlton, Study Director — Syntara
Locations (8):
- Australia (7):
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Childrens Hospital at Westmead, Sydney, New South Wales
  - Prince Charles Hospital, Brisbane, Queensland
  - Royal Children's Hospital, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
  - Sir Charles Gairdner, Perth, Western Australia
- Greenlane Hospital, Auckland, North Island, New Zealand

REFERENCES:
- [Result] Jaques A, Daviskas E, Turton JA, McKay K, Cooper P, Stirling RG, Robertson CF, Bye PTP, LeSouef PN, Shadbolt B, Anderson SD, Charlton B. Inhaled mannitol improves lung function in cystic fibrosis. Chest. 2008 Jun;133(6):1388-1396. doi: 10.1378/chest.07-2294. Epub 2008 Mar 13. PMID 18339790
- [Result] Daviskas E, Anderson SD, Jaques A, Charlton B. Inhaled mannitol improves the hydration and surface properties of sputum in patients with cystic fibrosis. Chest. 2010 Apr;137(4):861-8. doi: 10.1378/chest.09-2017. Epub 2009 Oct 31. PMID 19880909